CLINICAL TRIAL: NCT05585918
Title: R-CITY: A Collaborative Intervention With Teachers and Youth
Brief Title: The R-CITY Project: A Collaborative Intervention With Teachers and Youth
Acronym: R-CITY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Sheppard Pratt Health System (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Catherine Bradshaw, Professor; Senior Associate Dean for Research and Faculty Development, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBS2232
Record Dates: First submitted 2022-10-07; First posted 2022-10-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Violence

STUDY DESIGN:
Intervention Model Description: School-level randomization of teachers to arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Step Only (Active Comparator): Second Step Only Condition supports include:
  * School wide support for implementation of Second Step curriculum (e.g., technical assistance professional development, facilitated professional learning communities)
  * Support to Positive Behavioral Intervention and Supports (PBIS) and Multi Tiered System of Supports (MTSS) with alignment of initiatives
  * Individualized technical assistance with Second Step program implementation
  Interventions: Behavioral: Second Step Only
- Second Step + R-CITY (Experimental): Second Step + R-CITY supports include supports from the Second Step Only condition plus:
  * Training and implementation support for teachers to deliver 6 student lessons tailored to each grade level (4th and 5th for elementary schools; 6th - 8th for middle schools) and aligned with Second Step core content
  * Five 45-minute school-wide Professional Development (PD) sessions to complement the school district's PD
  * Individualized teacher coaching to support implementing teacher practices and classroom lessons
  Interventions: Behavioral: Second Step + R-CITY

INTERVENTIONS:
Behavioral: Second Step + R-CITY — For the Second Step + R-CITY (experimental) condition schools, activities include those in the Second Step Only condition, as well as student lessons designed by the project team, as well as training and individualized support for implementing classroom lessons, five 45-minute professional development sessions, and one-on-one coaching to support teacher practices and the implementation of the 6 classroom lessons.
  Other Names: R-CITY Intervention
  Arms: Second Step + R-CITY
Behavioral: Second Step Only — For the Second Step Only (active comparator) condition schools, activities involve school-wide technical assistance and implementation support for the Second Step program implementation, as well as individualized technical assistance for the Second Step program. In the year following participation, Second Step Only condition schools are offered access to and training and technical support for the classroom lessons.
  Arms: Second Step Only

SUMMARY:
"R-CITY" refers to the Collaborative Intervention with Teachers and Youth to practice and apply the 4 "Rs" of social skills in the classroom - Recognizing, Responding, Relationships, and Resilience. R-CITY is a collaborative teacher- and youth-focused prevention intervention that offers student lessons to accompany the Second Step curriculum. The lessons are designed to create safe and positive learning environments for all.

The R-CITY Project uses a school-level randomized controlled trial (RCT) design to test the integration of the Second Step program that the school district had been scaling up district wide with the R-CITY lessons. The purpose of the RCT is to determine the "value-added" of the Second Step program plus the new skill content compared to the Second Step alone in elementary and middle schools. Students in both conditions get access to the Second Step content, as an active control condition.

DETAILED DESCRIPTION:
The study aims to test the R-CITY intervention in 27 elementary and middle schools. Specific aims are as follows: Aim 1 is to test the effects of the integrated R-CITY intervention on attitudes. Aim 2 is to test the effects of the integrated R-CITY intervention on classroom practices and teaching self-efficacy. Aim 3 is to test the effects of the integrated R-CITY intervention on student behaviors. Outcomes are assessed at pre-test in the fall and post-test in the spring, over the course of the school year.

ELIGIBILITY:
Inclusion Criteria:

- General education teachers of core subjects (Mathematics, Science, Social Studies, English/Language Arts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
ASSIST Classroom Observations | Post-intervention, within one month following the completion of the intervention.
  The ASSIST is a direct observational measure that assesses the classroom interactions between students and teachers. Observation cycles are 15 minutes and scales include tallied counts of teacher and student behaviors, as well as global ratings of interactions based on a Likert-style scale.

SECONDARY OUTCOMES:
R-CITY Teacher Self-Report Survey | Post-intervention, within one month following the completion of the intervention.
  This survey assesses teachers' cultural competence and self-efficacy. Each item on this scale was scored on a 6-point Likert-type scale where 1 is strongly disagree and 6 is strongly agree.
Suspensions | Post-intervention, within one month following the completion of the intervention.
  School-level student suspensions (publicly reported and accessible).

CONTACTS AND LOCATIONS:
Locations (1):
- Shepard Pratt Health System, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT05585918/ICF_000.pdf